CLINICAL TRIAL: NCT05595512
Title: Risk Factors for Developing Maternal Postpartum Depression; A Retrospective Cross-sectional Study
Brief Title: Postpartum Depression
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Associate Professor, University of Jordan
Other Study IDs: JUH obstetrics
Record Dates: First submitted 2022-10-22; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Development of Depression Postpartum
Keywords: postpartum, depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Naser Al-Husban — depressive symptoms within 6 months of delivery

SUMMARY:
Postpartum depression (PPD) is one of the most common psychiatric complications of pregnancy and postpartum. It is often defined as an episode of depressive disorder that occurs in the postpartum period. Evidence suggests that PPD has serious consequences on the quality of life of all family members, increases the risk for familial conflicts, leaving great negative effects on maternal-infant interaction. The aim of our study was to investigate and shed the light on the determinants of development of PPD mainly maternal age among women in Jordan. We also aimed at examining additional factors on prevalence of PPD and providing more information on PPD among Jordanian mothers.

DETAILED DESCRIPTION:
This was a retrospective descriptive cross-sectional study and included patients were those diagnosed to have PPD within 6 months of delivery at Jordan University hospital (JUH) in the period 1st of January 2014 to the 1st of March 2021, Amman, Jordan. Data was collected retrospectively from the electronic files, from the departments of obstetrics and gynecology and psychiatry JUH in patients, outpatient clinics, inpatients' files delivery room records. All data are electronic in the period of the study. Inclusion criteria; patients with confirmed diagnosis of PPD with complete clinical data and have no other psychiatric diseases. Exclusion criteria; patients with maternal blues, patients with a diagnosis of any other psychiatric diseases, cases of unconfirmed depression and those with missing data.

Main outcome measure was the number of patients who developed PPD within 6 months of childbirth in relation to age, parity and mode of delivery. We collected data of patients who were confirmed to have a diagnosis of postpartum depression by a consultant psychiatrist in the hospital who followed diagnostic criteria of the American psychiatric association11. Intellectual disability was not specifically assessed in our patients.

The variables and information collected for this study included age, parity, mode of delivery, body mass index (BMI) that was objectively measured routinely in our obstetric population. In addition, medications, chronic diseases, past history of depression, psychiatry, breast feeding, and any social or marital problems were also retrieved. Data related to antenatal complications like antepartum hemorrhage (APH), diabetes mellitus (DM), preeclampsia toxemia (PET), urinary tract infection (UTI)/pyelonephritis necessitated hospital admission, postpartum hemorrhage (PPH) with no need for blood transfusion, PPH with blood transfusion, emergency hysterectomy for bleeding, fetal outcome including nursery (good, term), neonatal intensive care unit (NICU) admission: preterm, hypoxemia/acidosis, birth trauma, congenital anomalies, fetal loss [Intrauterine Fetal Death (IUFD), stillborn, neonatal] were also obtained

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed diagnosis of PPD
* with complete clinical data
* have no other psychiatric diseases

Exclusion Criteria:

* patients with maternal blues
* patients with a diagnosis of any other psychiatric diseases
* cases of unconfirmed depression
* those with missing data.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — more than 18 years of age and up to 49
Study Population: patients were those diagnosed to have PPD within 6 months of delivery at Jordan University hospital (JUH) in the period 1st of January 2014 to the 1st of March 2021, Amman, Jordan. Data was collected retrospectively from the electronic files, from the departments of obstetrics and gynecology and psychiatry JUH in patients, outpatient clinics, inpatients' files delivery room records
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Postpartum depression symptoms | 6 months
  symptoms related to depression that developed postpartum

IPD SHARING:
Plan to Share IPD: Undecided
available on reasonable request from the investigator